CLINICAL TRIAL: NCT05497687
Title: A Strength-building Lifestyle-integrated Intervention for Tackling Double Burden of Sarcopenic Patients With Coronary Artery Disease: A Pilot Randomized Controlled Trial
Brief Title: Strength-building Lifestyle-integrated Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Polly Wai-Chi Li, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UW22-516
Record Dates: First submitted 2022-08-03; First posted 2022-08-11 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Sarcopenia; Coronary Artery Disease
Keywords: cardiovascular disease; physical activity; sarcopenia; coronary artery disease; resistance exercise; older adults
MeSH Terms: conditions — Sarcopenia; Coronary Artery Disease; Cardiovascular Diseases; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Masked for the study arms allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 12-week strength-building intervention (Experimental): Participants in the intervention group will participate in a 12-week strength-building intervention comprising of face-to-face/remote sessions with telephone follow-ups.
  Interventions: Other: Resistance exercise
- Routine care that they currently receiving provided by their primary healthcare providers (No Intervention): The control group will receive routine care that they currently receiving provided by their primary healthcare providers, which include unstructured patient education on lifestyle modification. The usual care does not include structured exercise training.

INTERVENTIONS:
Other: Resistance exercise — The training schedule for supervised sessions (including community-based and home-based) will last for 60 minutes per session, two sessions per week. From Week 3 and 4, the exercise specialist will deliver supervised home-based training, with one in-person session via home visits and one session to be delivered remotely via an online platform (Zoom). Then the supervision will gradually tail off from Week 5 and onwards, from online supervised sessions, to unsupervised self-practice sessions. An in-person supervised home visit as a booster session will be given at Week 9, the beginning of the habituation phase. Telephone follow-ups will be arranged at Week 10 - 12 by the exercise specialist. All participants in the intervention group will be invited to take part in a qualitative interview to explore the feasibility and acceptability of the intervention.
  Arms: 12-week strength-building intervention

SUMMARY:
This study aims to 1) develop a strength-building lifestyle-integrated intervention for sarcopenic CAD patients and to 2) examine the feasibility and 3) preliminary effects of this intervention on skeletal muscle mass, muscle strength, physical performance, cardiac-related functional status and health-related quality of life (HRQoL), psychological distress, major adverse cardiovascular and cerebral events (MACCE) and hospital readmission rates

DETAILED DESCRIPTION:
Sarcopenia, a progressive and generalized skeletal muscle disorder characterized by accelerated loss of muscle mass and function, which is related to functional and physiological impairments.Individuals with sarcopenia are associated with profound adverse health outcomes, including increased incidents of falls and fractures, functional decline and increased all cause mortality. No study has been done to examine its effects on patients having the co-existence of sarcopenia and CAD, leaving a significant gap in the literature. Indeed, enabling this vulnerable cohort to adopt and maintain regular resistance exercise remains a great challenge. Assisting older adults to integrate exercise into daily activities can maximize the training benefits and overcome barriers to exercise, and thus improve exercise adoption and adherence. This study will include an assessor-blinded two-arm prospective pilot randomized controlled trial (RCT) and a qualitative study to determine the feasibility, acceptance and engagement experience of the participants in the strength-building lifestyle-integrated intervention with assessments measured at baseline, 3 months and 6 months after randomization. Patients will be allocated chronologically in a 1:1 ratio by using a computer-generated random sequence to determine the block size (4, 6 and 8) and respective study group allocation. Additional to the usual care provided by the primary healthcare providers (i.e. unstructured patient education on lifestyle modification without structured exercise training), the intervention group will participate in a 12-week strength-building intervention to be delivered by an exercise specialist who is required to have a Bachelor's degree in physical education, sports science, physiotherapy or equivalent, and at least 2 years of postgraduate experience.The control group will receive routine care that they currently receiving provided by their primary healthcare providers, which includes unstructured patient education on lifestyle modification. The usual care does not include structured exercise training. This study will be conducted in a patient mutual support organization Care for Your Heart. Muscle mass and strength, physical performance, cardiac-specific functional status, cardiac-specific HRQoL, psychological distress, MACCE and hospital readmission rate will be measured for outcome evaluation at baseline (T0), immediate postintervention (T1), and 3 months post-intervention (T2).Physical performance will be the primary outcome, while the remaining will be the secondary outcomes.

This study aims to 1) develop a strength-building lifestyle-integrated intervention for sarcopenic CAD patients and to 2) examine the feasibility and 3) preliminary effects of this intervention on skeletal muscle mass, muscle strength, physical performance, cardiac-related functional status and health-related quality of life (HRQoL), psychological distress, major adverse cardiovascular and cerebral events (MACCE) and hospital readmission rates.

The hypotheses for the first and third study aims are:

1. Patients with sarcopenia and coronary artery disease (CAD) receiving the intervention will present with increased skeletal muscle mass and strength compared with the control group at immediate post-intervention (T1), and 3 months post-intervention (T2).
2. Patients with sarcopenia and CAD receiving the intervention will present with improved physical performance, cardiac-related functional status, HRQoL and psychological distress compared to the control group at immediate postintervention (T1), and 3 months post-intervention (T2).
3. Patients with sarcopenia and CAD receiving the intervention will present with a lower rate of major adverse cardiovascular and cerebral events (MACCE) and hospital readmission compared to the control group at immediate post-intervention (T1), and 3 months post-intervention (T2).

The second aim is exploratory and qualitative, thus, there is no hypothesis to be tested.

ELIGIBILITY:
Inclusion Criteria:

* Chinese adults with a confirmed diagnosis of coronary artery disease (CAD);
* Age ≥60 years or older;
* Presence of sarcopenia according to the diagnostic criteria defined by the Asian Working Group for Sarcopenia1: low skeletal muscle mass (measuring the appendicular skeletal muscle mass with bioelectrical impedance analysis: <7.0 kg/m2 for men and <5.7 kg/m2 for women), accompanied by low muscle strength (handgrip strength <28 kg for men and <18 kg for women);
* Free from ischemic symptoms when performing activities of daily living;
* Living in the community.

Exclusion Criteria:

* Cannot read Chinese or with impaired cognition (Abbreviated Mental Test score ≤6) or communication;
* A pacemaker or implantable cardioverter defibrillator precluding the use of bioelectrical impedance analysis for body composition assessment;
* Physical limitations precluding exercise training, with any contraindication for exercise, any terminal or unstable conditions (e.g., malignant arrhythmia, severe aortic stenosis, cancer);
* Admitted or recently completed a structured cardiac rehabilitation program within the past 6 months

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Physical performance (measured by the Short Physical Performance Battery) | Changes from Baseline at the 3 months (after the intervention) and 6 months (follow-up)
  The Short Physical Performance Battery will be used to assess physical performance and is well validated and widely adopted in clinical and research settings. It is a brief performance-based assessment consisting of 3 timed-tasks, including standing balance, walking speed, and chair stand tests. The timed results will be rescaled to obtain a score ranging from 0 to 12, higher scores indicate better physical performance.

SECONDARY OUTCOMES:
Muscle mass | Changes from Baseline at the 3 months (after the intervention) and 6 months (follow-up)
  The appendicular skeletal muscle mass (ASM) will be measured with the bioelectrical impedance analysis (In-Body). This is one of the gold-standard evaluation tools suggested by international guidelines for assessment of muscle mass. It is widely used in research and hospital setting for clients with sarcopenia.
Muscle strength | Changes from Baseline at the 3 months (after the intervention) and 6 months (follow-up)
  The muscle strength will be measured with a hydraulic dynamometer ("Jamar" Dynamometer). The standard protocol suggested by international guidelines will be followed, the maximum reading of at least 2 trials using the dominant hand in a maximum-effort isometric contraction will be recorded.
Cardiac-specific functional status | Changes from Baseline at the 3 months (after the intervention) and 6 months (follow-up)
  The Seattle Angina Questionnaire will be used to measure cardiac-related functional status. It has 19 items in 5 subscales: physical limitation, angina stability, angina frequency, treatment satisfaction and disease perception. It is scored on a 1-5 or 6 sequentially coded scale and subscale scores are transformed to a scale of 0-100, with higher scores indicating higher levels of functioning and fewer limitations. The Chinese version has been shown to be reliable, valid, and sensitive to clinical change.
Cardiac-specific health-related quality of life (HRQoL) | Changes from Baseline at the 3 months (after the intervention) and 6 months (follow-up)
  The MacNew Heart Disease Health-related Quality of Life questionnaire (MacNew) will be used to measure cardiac-specific HRQoL. It has 27 items scored on a 1-7 scale, and then global score is calculated by summing the item scores, with higher scores representing better HRQoL. The global score ranges from 1 (low HRQoL) to 7 (high HRQoL). MacNew has good internal consistency, test-retest reliability, concurrent and discriminant validity.
Psychological distress | Changes from Baseline at the 3 months (after the intervention) and 6 months (follow-up)
  The Patient Health Questionnaire-4 (PHQ-4) will be used to measure psychological distress. It consists of 4 items assessing anxiety and depression, to be responded on a 4-point Likert scale. The composite total score ranges from 0 to 12, higher scores indicate greater level of anxiety and depression. It has good psychometric properties.
MACCE and hospital readmission rates | Changes from Baseline at the 3 months (after the intervention) and 6 months (follow-up)
  Major adverse cardiovascular and cerebral events (MACCE) and hospital readmission rates.

CONTACTS AND LOCATIONS:
Overall Officials: Polly Li, Dr, Principal Investigator — The University of Hong Kong, School of Nursing
Locations (1):
- The School of Nursing, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Li PWC, Yu DSF, Chan NY, Chiu SH, Leung JYH, Ye EQH, Cheng MHK. Resistance-based exercise intervention for patients with coronary artery disease and sarcopenia: a pilot randomized controlled trial. Eur J Cardiovasc Nurs. 2025 Jul 21;24(5):736-745. doi: 10.1093/eurjcn/zvaf041. PMID 40114426

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-30): https://cdn.clinicaltrials.gov/large-docs/87/NCT05497687/Prot_SAP_000.pdf